CLINICAL TRIAL: NCT02201732
Title: Assessment of the Effectiveness of Hysteroscopy in the Treatment of Intrauterine Trophoblastic Retentions
Brief Title: Effectiveness of Hysteroscopy in the Treatment of Intrauterine Trophoblastic Retentions
Acronym: HY-PER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P130920; 2014-A00340-47
Record Dates: First submitted 2014-07-17; First posted 2014-07-28 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Incomplete Miscarriage
Keywords: Incomplete miscarriage; Hysteroscopy; curettage, pregnancy; RCT
MeSH Terms: conditions — Abortion, Incomplete | interventions — Hysteroscopy; Curettage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A : Operative hysteroscopy (Experimental): operative hysteroscopy with direct visualization
  Interventions: Procedure: Hysteroscopy
- Arm B : Aspirative curettage (Active Comparator): curettage is the standard surgical treatment in most centers
  Interventions: Procedure: Curettage

INTERVENTIONS:
Procedure: Hysteroscopy — Performed under general or local anesthesia, antibioprophylaxis in accordance to center practices may be administered. Cervical dilatation, will be made in order to introduce the hysteroscope. Operative hysteroscope used will include a handle. The distension of the uterine cavity will be performed with physiological saline or glycocoll, depending on the polarity of the high frequency generator necessary for resection system (monopolar or bipolar), with a pressure of maximum irrigation of 110 mm Hg.
  Arms: Arm A : Operative hysteroscopy
Procedure: Curettage — Performed under general or local anesthesia, the used material may be rigid or flexible vacurette. In the same way, the prophylactic antibiotic, the diameter of the used vacurette, the importance of cervical dilation necessary and a possible peroperative ultrasound guidance will be left at the discretion of the operator and habits of the center. A check of the uterine vacuity by foam curette will be conducted at the end of curettage.
  Arms: Arm B : Aspirative curettage

SUMMARY:
The purpose of this study of is to compare subsequent fertility rates between hysteroscopy and aspirative curettage in the surgical treatment of incomplete spontaneous abortion

DETAILED DESCRIPTION:
Incomplete spontaneous abortion (ISA) is defined by the intrauterine retention of conceptual product after incomplete or partial expulsion of the conceptual product. Treatment such retention may be expectant care, medical treatment or surgery. Currently, curettage is the standard surgical treatment in most centers. However, operative hysteroscopy, in addition to the direct visualization of the retained conceptual product, in contrast to the curettage, would allow elective evacuation of retention while reducing surgical complications. Studies of low effective, retrospective, have found an fertility's increase in patients treated by operative hysteroscopy. These data need to be confirmed by a randomized controlled trial in order to change the standard surgical treatment of this disease if hysteroscopy procedure would found to be superior.

We propose a multicenter - single blind - randomized - therapeutic study. Randomization will concern the surgical procedure in patients treated surgically for intrauterine retention after spontaneous miscarriage. Randomization will be performed at the admission to the patient in the operating room by electronic means using a secure internet platform, single-blind for the patient with unblinding at the end of the trial or in case of complication. The patient will be randomly assigned to one of two treatment arms following:

* Arm A : Operative hysteroscopy
* Arm B : Aspirative curettage The inclusion will be performed at time of diagnosis (incomplete miscarriage) with an ultrasound of intrauterine retention for which surgical treatment has been decided. The initial medical examination (inclusion visit) will include a complete gynecological examination. The diagnosis of incomplete miscarriage will be performed using a transvaginal pelvic ultrasound. Transvaginal ultrasound will be performed according to a technique of standardized pelvic ultrasound ; the retention will be diagnosed in the presence of a heterogeneous image or intrauterine gestational sac more than 15 mm in thickness. On this visit, the patient will complete a questionnaire concerning her medical histories and the aborted pregnancy.

Patients will have a care in accordance with center practices for the hospital stay. Surgical treatment will be performed within the time depending on the availability of the operating room of participating center.

A hospitalization report indicating the participation to the study, but not mentioning the treatment group, will be sent to the attending physician and the patient. An information form with postoperative instructions will be given to patients included in this protocol without mentioning the surgical arm. The operative report will be given to the patient at the end of her participation in the trial.

A total of five visits (including final visit) are scheduled for this trial. The patient will be monitored in the form of telephone conversation or questionnaire sent by email or post. Monitoring will be done by the investigator that enrolled the patient with the help of the URC in charge of the project. In case of complications, failure of the intervention or diagnosis of a uterine cavity pathology, the care will be left to the discretion of the medical center team.

ELIGIBILITY:
Inclusion Criteria:

* Major, under 45 years with intrauterine trophoblastic retention after incomplete miscarriage in the first quarter (termination of pregnancy < 14 WA),
* With desire of pregnancy ;
* Intrauterine trophoblastic retention diagnosed by transvaginal pelvic ultrasound finding a intrauterine heterogeneous image or intrauterine gestational sac more than 15 mm in thickness, complicated or not of endometritis ;
* Decision to surgical management of incomplete miscarriage by the health care team ;
* Patient beneficiary or affiliated to a health insurance
* Informed and signed consent

Exclusion Criteria:

Will not be included in the protocol patients :

* having a uterine malformation known ;
* having received surgical treatment for the current intrauterine retention ;
* with intrauterine retention diagnosed by transvaginal pelvic ultrasound of more than 50 mm in thickness ;
* requiring a haemostatic act in urgency for heavy vaginal bleeding (miscarriage haemorrhage) ;
* bearer of intrauterine device ;
* having an evolutive pregnancy;
* having an ectopic pregnancy;
* having a trophoblastic retention following a voluntary abortion ;
* having a pregnancy achieved by medically assisted procreation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 577 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Progressive intrauterine pregnancy > 22 WA | Until 2 years post surgery
  Questionnaire

SECONDARY OUTCOMES:
Next pregnancy | Until 2 years post surgery
Surgical complications' rate | until 2 years post surgery
  Clavien-Dindo classification
Surgical reinterventions | until 2 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud FAUCONNIER, MD, PhD, Study Director — Centre Hospitalier Intercommunal de Poissy / Saint-Germain
Locations (1):
- Centre hospitalier intercommunal de poissy-saint germain en Laye, Poissy, France

REFERENCES:
- [Background] Huchon C, Drioueche H, Koskas M, Agostini A, Bauville E, Bourdel N, Fernandez H, Fritel X, Graesslin O, Legendre G, Lucot JP, Panel P, Raiffort C, Giraudet G, Bussieres L, Fauconnier A. Operative Hysteroscopy vs Vacuum Aspiration for Incomplete Spontaneous Abortion: A Randomized Clinical Trial. JAMA. 2023 Apr 11;329(14):1197-1205. doi: 10.1001/jama.2023.3415. PMID 37039805
- [Background] Huchon C, Koskas M, Agostini A, Akladios C, Alouini S, Bauville E, Bourdel N, Fernandez H, Fritel X, Graesslin O, Legendre G, Lucot JP, Matheron I, Panel P, Raiffort C, Fauconnier A. Operative hysteroscopy versus vacuum aspiration for incomplete spontaneous abortion (HY-PER): study protocol for a randomized controlled trial. Trials. 2015 Aug 19;16:363. doi: 10.1186/s13063-015-0900-1. PMID 26282937
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352